CLINICAL TRIAL: NCT01521390
Title: Randomized, Double-blind, 5 Period Cross Over Study Assessing Lung Function in Healthy Volunteers Following Single Inhalations of GSK573719 Inhalation Powder From Two Configurations of the Novel Dry Powder Inhaler
Brief Title: Assessment of Lung Function After Single Inhalations of a Bronchodilator From 2 Configurations a Dry Powder Inhaler.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 115487
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Other): Subjects receive one inhalation from each intervention
  Interventions: Drug: GSK573719 62.5 mcg (one strip); Drug: GSK573719 62.5 mcg(two strips); Drug: GSK573719 125 mcg (one strip); Drug: GSK573719 125 mcg(two strips); Drug: Placebo

INTERVENTIONS:
Drug: GSK573719 62.5 mcg (one strip) — GSK573719 62.5 mcg delivered by 1 strip configuration of novel dry powder inhaler
Drug: GSK573719 62.5 mcg(two strips) — GSK573719 62.5 mcg delivered by 2 strip configuration of novel dry powder inhaler
Drug: GSK573719 125 mcg (one strip) — GSK573719 125 mcg delivered by 1 strip configuration of novel dry powder inhaler
Drug: GSK573719 125 mcg(two strips) — GSK573719 125 mcg delivered by 2 strip configuration of novel dry powder inhaler
Drug: Placebo — Placebo, no active ingredient

SUMMARY:
GSK573719 is a high-affinity specific muscarinic receptor (mAChR) antagonist which is being developed for the treatment of chronic obstructive pulmonary disease (COPD). The long duration of action of GSK573719, when administered via inhalation to humans supports the potential for use as a long acting bronchodilator.This is a randomized, double-blind, placebo-controlled, 5 period cross-over study in healthy male and female volunteers. The study will measure lung function after single inhaled doses from two configurations of the Novel Dry Powder Inhaler. Key assessments will include clinical relevant PD parameters: sGaw, FEV1

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy male or female as determined by a responsible and experienced physician, based on a medical evaluation including [medical history, physical examination, laboratory tests and cardiac monitoring]. A subject with a clinical significant abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator believes that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.]
  * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 10 days after last dose.
* Body weight ≥ 50 kg and BMI within the range 19.0 - 29.9 kg/m2 (inclusive).
* Normal spirometry (FEV1 ≥ 80% of predicted, FEV1/FVC ≥ 70%).
* Response to ipratropium bromide defined as

  * an increase in sGaw of ≥25% over pre-dose baseline at 2 h following 80μg ipratropium bromide; or
  * a documented increase in sGaw of ≥25% over pre-dose baseline at 2 h following inhalation of 80 μg of ipratropium bromide within 3 months of screening.
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* No significant abnormality on 12-lead ECG at screening, including QTcF < 450msec.
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked))
* Subjects who are able to use the Novel DPI satisfactorily
* Subjects, who are capable of giving written informed consent, have signed and dated the informed consent form which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A supine mean heart rate outside the range 40-90 beats per minute (BPM) at screening.
* A supine blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHG) at screening.
* History of symptomatic arrhythmias.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

  • an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Subject who has asthma or a history of asthma or bronchoconstriction.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco or nicotine-containing products within 6 months prior to screening.
* Subjects who are kept due to regulatory or juridical order in an institution.
* Subjects who are in military service.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-10-12 (Actual); Primary Completion 2011-12-16 (Actual); Study Completion 2011-12-16 (Actual)

PRIMARY OUTCOMES:
Weighted mean and maximal change from baseline in sGaw | serial over 24 hr for each treatment period
  measured by plethysmography, for each inhaled dose from one strip configuration as compared with two strip

SECONDARY OUTCOMES:
Plasma concentration of GSK573714 | over 24 hrs for each treatment period
  Pharmacokinetic parameters
Urine concentration of GSK573714 | over 24 hr for each treatment period
  Pharmacokinetic parameters
Blood pressure | over 24 hr for each treatment period
Heart Rate | over 24 hr for each treatment period
Serial FEV1 | over 24 hr
Serial sGaw | over 24 hr for each treatment period
ECG | over 24 hrs for each treatment period
  12-lead ECG
Clinical lab safety tests | Over 24 hrs for each treatment period
  Haematology, Biochemistry and Urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115487 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115487?search=study&search_terms=115487#rs
- Available data/document: Individual Participant Data Set: 115487 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115487 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115487 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115487 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115487 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115487 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115487 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register